CLINICAL TRIAL: NCT03043053
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effects of Repeat Doses of Intranasal Oxytocin in Obese Adults
Brief Title: The Effects of Oxytocin in Obese Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Elizabeth Austen Lawson, Associate Professor of Medicine, Harvard Medical School, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016P002810
Record Dates: First submitted 2017-02-01; First posted 2017-02-03 (Estimated); Results first posted 2024-02-07 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2024-01

CONDITIONS: Obesity
Keywords: weight loss; body mass index; oxytocin; magnetic resonance imaging
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- oxytocin (Experimental): oxytocin nasal spray (24 IU nasal spray, 4 times per day for 8 weeks)
  Interventions: Drug: oxytocin nasal spray
- placebo (Placebo Comparator): placebo nasal spray (4 times per day for 8 weeks)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: oxytocin nasal spray — oxytocin intranasal spray
  Other Names: Syntocinon
  Arms: oxytocin
Drug: Placebo — Placebo nasal spray
  Arms: placebo

SUMMARY:
This is a randomized, double blind, placebo-controlled study of the effects of intranasal oxytocin in obese adults, ages 18-45 years old. Subjects will be randomized to receive of intranasal oxytocin or placebo (3 sprays per nostril, 4 times per day) for 8 weeks. Study visits include screening to determine eligibility, a 2-part baseline visit, and visits every 2 weeks thereafter until week 14, with a safety follow-up visit 6 weeks after the last dose of study drug. Study procedures include behavioral, metabolic, neuroimaging, and endocrine assessments.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old;
* BMI greater than or equal to 30 kg/m2

Exclusion Criteria:

* Use of drug affecting metabolism, glucose, or appetite (Metformin is allowed if dose and weight are stable for at least 3 months);
* history of medication changes within 4 weeks of enrollment;
* active substance use;
* history of cardiovascular disease, gastrointestinal disorders, bariatric surgery, epilepsy, untreated thyroid disease;
* hematocrit >2% below normal;
* fasting glucose > 125 mg/dL or hemoglobin A1c ≥ 7% ;
* ALT or AST >2.5 times upper limit of normal;
* Cr >1.5 mg/dL; hyponatremia;
* pregnancy or breastfeeding;
* unwilling to use medically acceptable form of contraception (females only)
* follows a nonstandard diet (e.g., gluten free, pescatarian, vegetarian, vegan, Paleo, Atkins, raw diet, macrobiotic diet)
* current smoking or tobacco use

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2022-05-20 (Actual); Study Completion 2022-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Lawson, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Plessow F, Kerem L, Wronski ML, Asanza E, O'Donoghue ML, Stanford FC, Eddy KT, Holmes TM, Misra M, Thomas JJ, Galbiati F, Muhammed M, Sella AC, Hauser K, Smith SE, Holman K, Gydus J, Aulinas A, Vangel M, Healy B, Kheterpal A, Torriani M, Holsen LM, Bredella MA, Lawson EA. Intranasal Oxytocin for Obesity. NEJM Evid. 2024 May;3(5):EVIDoa2300349. doi: 10.1056/EVIDoa2300349. Epub 2024 Apr 23. PMID 38815173

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oxytocin | Placebo
Started (Safety cohort includes all randomly assigned participants who received at least one dose of study drug) | 31 | 30
Started (mITT) (Modified Intention-To-Treat (mITT) cohort is defined as all subjects who completed at least 1 visit while on study drug) | 31 | 29
Completed (Completed cohort (safety and mITT) includes all randomly assigned participants who received at least one dose of study drug and completed the study to Week 14) | 28 | 22
Not Completed | 3 | 8

BASELINE CHARACTERISTICS:
Population: Safety cohort, which was defined as all randomly assigned participants who received at least one dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxytocin | Placebo | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (6.1) | 33.2 (6.4) | 33.6 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 33
  Male | 14 | 14 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 25 | 23 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 3 | 13
  White | 15 | 23 | 38
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Mean Difference in Weight Loss Between Oxytocin and Placebo 8 Weeks After Baseline
Description: The mean difference in weight loss between oxytocin- and placebo-treated groups from baseline to 8 weeks. All participants of the modified intention-to-treat cohort were aggregated into a single linear mixed effects model with the factors Time (Baseline, Week 2, Week 4, Week 6, and Week 8) and Group (oxytocin/placebo) and the interaction Time*Group controlled for sex (male/female) and obesity class (class I, II, and III) to produce a single value (estimated mean difference) and 95% confidence interval for the difference between groups and a single value (estimated mean change) within each group.
Time Frame: Baseline to 8 weeks
Population: Modified Intention-To-Treat cohort, which includes all randomly assigned participants who completed at least 1 visit on study drug.
Measure: Number; unit: kilogram
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 31 | 29
kilogram | 0.20 | 0.26
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Other; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-1.4 to 1.3]

2. Secondary Outcome: Change in Resting Energy Expenditure After 8 Weeks of Oxytocin Versus Placebo
Description: The mean difference in resting energy expenditure between oxytocin- and placebo-treated groups from baseline to 8 weeks. All participants of the modified intention-to-treat cohort were aggregated into a single linear mixed effects model with the factors Time (Baseline and Week 8) and Group (oxytocin/placebo) and the interaction Time*Group controlled for sex (male/female), obesity class (class I, II, and III), and lean mass to produce a single value (estimated mean difference) and 95% confidence interval for the difference between groups and a single value (estimated mean change) within each group. Reported are model estimates rounded to one decimal.
Time Frame: Baseline to 8 weeks
Population: as for outcome 1
Measure: Number; unit: kilocalories/day
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 31 | 29
kilocalories/day | -17.8 | 11.8
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Other; Mean Difference (Final Values) = -29.7, 95% CI 2-sided [-141.9 to 82.6] — Controlled for lean mass. Reported values are outputted by STATA

3. Secondary Outcome: Change in Fat Depots After 8 Weeks of Oxytocin Versus Placebo
Description: The mean difference in total fat mass between oxytocin- and placebo-treated groups from baseline to 8 weeks. All participants of the modified intention-to-treat cohort were aggregated into a single linear mixed effects model with the factors Time (Baseline and Week 8) and Group (oxytocin/placebo) and the interaction Time*Group controlled for sex (male/female) and obesity class (class I, II, and III) to produce a single value (estimated mean difference) and 95% confidence interval for the difference between groups and a single value (estimated mean change) within each group.
Time Frame: Baseline to 8 weeks
Population: as for outcome 1
Measure: Number; unit: gram
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 31 | 29
gram | 248.5 | 52.5
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Other; Mean Difference (Final Values) = 196.0, 95% CI 2-sided [-1036 to 1428]

4. Secondary Outcome: Difference in Caloric Intake After 6 Weeks of Oxytocin Versus Placebo
Description: The mean difference in caloric intake between oxytocin- and placebo-treated groups from baseline to 6 weeks. All participants of the modified intention-to-treat cohort were aggregated into a single linear mixed effects model with the factors Time (Baseline and Week 6) and Group (oxytocin/placebo) and the interaction Time*Group controlled for sex (male/female) and obesity class (class I, II, and III) to produce a single value (estimated mean difference) and 95% confidence interval for the difference between groups and a single value (estimated mean change) within each group.
Time Frame: Baseline to 6 weeks
Population: as for outcome 1
Measure: Number; unit: kilocalories
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 31 | 29
kilocalories | -31.4 | 120.6
Statistical Analysis 1: Comparison: Oxytocin vs Placebo; Test type: Other; Mean Difference (Final Values) = -152.0, 95% CI 2-sided [-302.3 to -1.7]

ADVERSE EVENTS:
Time Frame: Baseline to Week 14 end of study
Description: Adverse events and serious adverse events reported are those that started or worsened after the first dose of study treatment to the end of the study at Week 14.
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 24/31 | 23/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oxytocin (N=31) | Placebo (N=30)
Ventricular arrhythmia (Cardiac disorders) | 0 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distention (Gastrointestinal disorders) | 0 | 1
Abdominal tenderness (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 2
Chest pain (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 2
Gastrointestinal viral infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 2
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 4 | 3
Blood potassium decreased (Investigations) | 0 | 1
Blood potassium increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 1 | 0
Blood sodium decreased (Investigations) | 0 | 1
Liver function test increased (Investigations) | 2 | 3
Gout (Metabolism and nutrition disorders) | 0 | 1
Polydipsia (Metabolism and nutrition disorders) | 0 | 1
Thirst (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 5 | 7
Parasthesia (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Dysphoria (Psychiatric disorders) | 1 | 2
Hypersomnia (Psychiatric disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Polyuria (Renal and urinary disorders) | 1 | 0
Uterine pain (Reproductive system and breast disorders) | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acne (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 2
Skin infection (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Wound complication (Skin and subcutaneous tissue disorders) | 2 | 0
Hypertension (Vascular disorders) | 1 | 2
Presyncope (Vascular disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-07): https://cdn.clinicaltrials.gov/large-docs/53/NCT03043053/Prot_SAP_000.pdf